CLINICAL TRIAL: NCT00617981
Title: A Phase III, Randomized, Double-Blinded, Dummy-Controlled Study of the Efficacy and Safety of ThermoDox® (Thermally Sensitive Liposomal Doxorubicin) in Combination With Radiofrequency Ablation (RFA) Compared to RFA-Alone in the Treatment of Non-Resectable Hepatocellular Carcinoma
Brief Title: Phase 3 Study of ThermoDox With Radiofrequency Ablation (RFA) in Treatment of Hepatocellular Carcinoma (HCC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Imunon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 104-06-301
Record Dates: First submitted 2008-02-06; First posted 2008-02-18 (Estimated); Results first posted 2017-03-24 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; liver cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ThermoDox + RFA (Experimental): ThermoDox 50 mg/m2 start infusion over 30 minutes about 15 minutes before radiofrequency ablation begins.
  Interventions: Drug: ThermoDox
- Sham + RFA (Sham Comparator): Sham infusion over 30 minutes about 15 minutes before radiofrequency ablation begins.
  Interventions: Drug: 5% Dextrose Solution

INTERVENTIONS:
Drug: ThermoDox — Thermally Sensitive Liposomal Doxorubicin 50 mg/m2 Single 30 minute intravenous infusion
  Arms: ThermoDox + RFA
Drug: 5% Dextrose Solution — Single 30 minute intravenous infusion
  Arms: Sham + RFA

SUMMARY:
The purpose of this study is to determine whether ThermoDox, a thermally sensitive liposomal doxorubicin, is effective in the treatment of non-resectable hepatocellular carcinoma when used in conjunction with radiofrequency ablation (RFA).

DETAILED DESCRIPTION:
This will be a Phase III, randomized, double-blinded, dummy-controlled, efficacy, and safety study of ThermoDox plus RFA versus RFA plus dummy infusion.

The 50 mg/m2 ThermoDox or dummy infusion will be administered IV over 30 minutes. As part of blinded pre-medication ThermoDox treated subjects will receive 20 mg of dexamethasone orally 48 hours prior to the drug infusion for infusion reaction prophylaxis. Subjects on the control arm will receive a matching dummy pre-medication pill orally at 48 hours prior to infusion of the study treatment. Thirty minutes prior to receiving the ThermoDox infusion, subjects will receive a blinded dose of 20 mg of IV dexamethasone, 50 mg IV diphenhydramine and either 50 mg of IV ranitidine or 20 mg of IV famotidine. Subjects on the control arm will receive a masked dummy pre-medication pill orally at 48 hours prior to infusion of the study medication, and a dummy infusion 30 minutes prior to dummy infusion of D5W (250 cc of 5% Dextrose solution). RFA will be initiated approximately at a minimum of 15 minutes after the initiation of study drug infusion and should be completed no later than 3 hours after study drug infusion initiation. The total length of the RFA procedure is proportional to the size of the tumor(s) involved and is anticipated to range from 12 to 60 minutes for each lesion with an estimated overall procedure time of less than 3 hours.

Subjects with incomplete ablations will be re-treated to complete the ablation according to the treatment assigned at randomization. The completion of an ablation in this manner will restart the timeline of the study-related visits/procedures. This repeated ablation procedure cannot occur earlier than 21 days post-ablation but no later than 14 days after the first post-ablation CT scan assessment. These subjects will start over at screening (see Table 1). If a complete ablation is not achieved after these two study treatments, the subject will be considered a treatment failure and the patient will be discontinued and followed for survival only.

Subjects who recur with local and/or distant intrahepatic HCC after a complete initial ablation will have met the primary endpoint of progression-free survival. However, if these subjects have lesions that are amenable to RFA the standard of care is to consider them for repeat RFA. Therefore, these subjects may receive treatment to which they were randomized if they continue to meet the inclusion and exclusion criteria of the protocol. Subjects who develop any extrahepatic lesion will have met the primary endpoint and will be discontinued from study treatment but will still be followed for overall survival.

Dynamic Contrast CT imaging will be used to assess the effectiveness of the ablation therapy. The blind will be maintained at the level of CT scan reads. All protocol-specified CT images will be centrally read and assessed by the endpoint committee in a blinded fashion. Posttreatment CT scans will be obtained at months 1, 3, 5, 7, 9 and 12 and every three months thereafter until withdrawal. Adverse event assessments and laboratory examinations will occur at each visit. All subjects will be monitored throughout the investigational period.

Patients that meet inclusion/exclusion criteria may be at risk for contrast-induced nephropathy (CIN) when undergoing the required CT with contrast procedures. The investigators must be mindful of the risk factors (e.g. diabetes, borderline renal function) associated with CIN and employ strategies to reduce the risk of CIN. In subjects with diabetes or borderline renal function (creatinine greater than 1.5 mg/dL) special precautions (e.g. hydration, contrast dose reduction, follow up creatinine determination) should be employed. An accepted procedure is adequate intravenous volume expansion with isotonic saline (1.0 - 1.5 mL/kg per hour) for 3-12 hours before the procedure and continued for 6-24 hours.

All randomized subjects will be followed for safety and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed hepatocellular carcinoma (HCC)
* No more than 4 HCC lesions with at least one ≥ 3.0 cm and none > 7.0 cm in maximum diameter, based on diagnosis at screening.
* If a subject has a large lesion (5.0 - 7.0 cm), any other lesions must be less than 5.0 cm.
* Anticipated ablation volume will be no larger than either removal of 3 hepatic segments or removal of more than 30% of total liver volume (as per maximum surgical limit).
* If additional lesions are discovered during the laparoscopic or open treatment procedure, that were undetectable by CT at screening, the size and location of the lesion(s) will be recorded in the CRF and the lesions will be treated at the discretion of the physician and guided by the local standard of care. The subject will remain on study if all lesions are treated. If any lesions cannot be completely ablated within two treatment attempts the subject will be considered a treatment failure.
* Study subjects being considered for re-treatment after disease progression may have more than 4 lesions.
* Male or female 18 years of age or older.
* Are willing to sign an informed consent form, indicating that they are aware of the investigational nature of this study that is in keeping with the policies of the institution.
* Be an appropriate candidate for receiving RFA as a medically indicated treatment as evaluated by the following factors:

  * Number of lesions
  * Size of lesions
  * Overall health of liver
  * Not a candidate for surgical resection
* Have an echocardiogram revealing a Left Ventricular Ejection Fraction (LVEF) ≥ 50%. Measurements with a multiple gated acquisition (MUGA) scan are allowed if an echocardiogram cannot be performed. The same method of measurement should be used to evaluate ejection fraction (EF) of the subject for the duration of the study.
* Willing to return to the study site for their study visits.
* Have life expectancy of ≥ 4 months.
* Have Child-Pugh Class A or B liver disease without encephalopathy or/and ascites.

Exclusion Criteria:

* Have serious medical illnesses including, but not limited to, congestive heart failure, myocardial infarction or cerebral vascular accident within the last six months, or life threatening cardiac arrhythmias.
* Is scheduled for liver transplantation.
* Have previously received any treatment for HCC (except for study subjects being considered for completion of treatment or re-treatment).
* Have previously received any doxorubicin (study subjects being considered for completion of treatment or re-treatment may have received ThermoDox previously).
* Have extrahepatic metastasis.
* Are pregnant or breast-feeding. In women of childbearing potential, a negative pregnancy test (serum) is required prior to study treatment.
* Women of childbearing potential who are not practicing an acceptable form of birth control (i.e. diaphragm, cervical cap, condom, surgical sterility or birth control pills. Women whose partner has undergone a vasectomy must use a second form of birth control).
* Have any known allergic reactions to any of the drugs or liposomal components or intravenous imaging agents to be used in this study.
* Have portal or hepatic vein tumor invasion/thrombosis.
* Have INR > 1.5 times the institution's upper normal limit (UNL), except in subjects who are therapeutically anticoagulated for medical conditions unrelated to HCC such as atrial fibrillation. Subjects may be re-screened after condition is treated or anticoagulant is withheld.
* Have platelet count < 75,000/mm3, absolute neutrophil count < 1500/mm3, or Hgb < 10.0 g/dL (unless the hemoglobin value has been stable, the subject is cardiovascularly stable, asymptomatic and judged able to withstand the RFA procedure).
* Have serum creatinine ≥ 2.5 mg/dL or calculated creatinine clearance (CrCl) ≤ 25.0 mL/min.
* Have serum bilirubin > 3.0 mg/dL.
* Have serum albumin < 2.8 g/dL.
* Have body temperature >1010F (38.30C) immediately prior to study treatment.
* Have contraindications to receiving doxorubicin HCl.
* Are being treated with other investigational agents.
* Use of an investigational drug within 30 days or 5 half-lives, whichever is longer, preceding the first dose of study medication (study subjects being considered for completion of treatment or re-treatment may have received ThermoDox previously).
* Have other concurrent malignancy (subjects with treated squamous cell carcinoma of the skin or basal cell carcinoma of the skin may be included), evidence of extrahepatic cancer from their primary malignancy, or ongoing, medically significant active infection.
* Documented HIV positive.
* NYHA class III or IV functional classification for heart failure.
* Evidence of hemachromatosis.
* Have history of contrast-induced nephropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 701 (Actual)
Dates: Start 2008-05 (Actual); Primary Completion 2013-01 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronnie T Poon, M.D., Study Director — Queen Mary Hospital, University of Hong Kong; Riccardo Lencioni, M.D., Study Director — University of Pisa
Locations (79):
- United States (9):
  - UCLA, Los Angeles, California
  - Mayo Clinic - Jacksonville, Florida, Jacksonville, Florida
  - University Of Louisville, Louisville, Kentucky
  - Mayo Clinic, Rochester, Minnesota
  - Mount Sinai School of Medicine, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Geisinger Health System, Wilkes-Barre, Pennsylvania
  - University of Texas Health Science Center, San Antonio, Texas
- Canada (2):
  - Vancouver General Hospital, Vancouver, British Columbia
  - Toronto General Hospital, Toronto, Ontario
- China (16):
  - The 1st Affiliated Hospital, Fujian Medical University, Fuzhou, Fujian
  - Tongji Hospital, Wuhan, Hubei
  - Nanjing Drum Tower Hospital, The Affilitated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - The First Affiliated Hospital of Suzhou University, Suzhou, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing
  - Beijing Cancer Hospital, Peking University School of Oncology, Beijing
  - Beijing You An Hospital, Capital Medical University, Beijing
  - Beijing You An Hospital，Capital Medical University, Beijing
  - Southwest Hospital, The First Affiliated Hospital of the Third Military Medical University, Chongqing
  - Sun Yat-Sen University Cancer Center, Guangzhou
  - Oncology Center of Nanfang Hospital, Southern Medical University, Guangzhou
  - Shanghai Changhai Hospital, Second Military Medical University, Shanghai
  - Tianjin No. 3 Central Hospital, Tianjin
- Queen Mary Hospital, Hong Kong, Hong Kong
- Italy (8):
  - Azienda Ospedaliera di Padova, Padua, Veneto
  - Azienda Ospedaliero-Universitaria di Bologna Policlinico S.Orsola Malpighi, Bologna
  - Ospedale Classificato San Giuseppe, Milano, Milan
  - Azienda Ospedaliera San Gerardo, Monza
  - Istituto Nazionale per lo Studio e la Cura dei Tumori "Fondazione Pascale" di Napoli, Napoli
  - Azienda Ospedaliero-Univeristaria Pisana, Pisa
  - Istituto dei Tumori Regina Elena, Roma
  - Azienda Sanitaria Ospedaliera Ordine Mauriziano di Torino Presidio Ospedaliero "Umberto I", Torino
- Japan (13):
  - Chiba University Hospital, Chiba
  - Yamanashi Prefectural Central Hospital, Kofu
  - Mie University Hospital, Mie
  - Saiseikai Niigata Daini Hospital, Niigata
  - Okayama University Hospital, Okayama
  - Iwate Medical University Hospital, Shiwa
  - Kyoundo Hospital, Tokyo
  - The University of Tokyo Hospital, Tokyo
  - Japanese Red Cross Medical Center, Tokyo
  - JR Tokyo General Hospital, Tokyo
  - Kanto Central Hospital, Tokyo
  - Wakayama Medical University, Wakayama
  - Yokohama City University Medical Center, Yokohama
- University Malaya Medical Centre, Kuala Lumpur, Malaysia
- Philippines (4):
  - Chinese General Hospital and Medical Center, Santa Cruz, Manila
  - The Medical City, Pasig, National Capital Region
  - St. Luke's Medical Center, Quezon City
  - Cardinal Santos Medical Center, San Juan City
- South Korea (12):
  - Soonchunhyang University Bucheon Hospital, Gyeonggi-do, Bucheon-si
  - Samsung Medical Center, Seoul, Gangnam-gu
  - Inje University Ilsan Paik Hospital, Gyeonggi-do, Goyang-si
  - Kyungpook National University Hospital, Daegu, Gyeongsangbuk-do
  - Seoul National University Hospital, Seoul, Jongno-gu
  - Kyungpook National University Hospital, Daegu, Jung-gu
  - The Catholic University of Korea, Kangnam St.Mary's Hospital, Seoul, Seocho-gu
  - Pusan National University Hospital, Busan
  - Seoul National University Bundang Hospital, Seongnam-si
  - Yonsei University Severance Hospital, Seoul
  - Korea University Medical Center Anam Hospital, Seoul
  - Asan Medical Center, Seoul
- Taiwan (9):
  - Chang Gung Memorial Hospital - Kao Shiung, Niaosong, Kaohsiung County
  - Chang Gung Memorial Hospital - Linkou, Linkou District, Taoyuan
  - Chang-Gung Memorial Hospital - Chiayi Branch, Chiayi City
  - Chang Gung Memorial Hospital - Keelung, Keelung
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
- Thailand (4):
  - Songklanagarind Hospital, Hat Yai, Changwat Songkhla
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Thammasat University Hospital, Pathum Thani

RESULTS

PARTICIPANT FLOW:
Groups:
- ThermoDox + RFA: ThermoDox should be administered at 50 mg/m2. The infusion should start approximately 15 minutes before radiofrequency ablation begins and continue for approximately 30 minutes.
  ThermoDox: Thermally Sensitive Liposomal Doxorubicin 50 mg/m2 Single 30 minute intravenous infusion
- Sham + RFA: Sham infusion should start approximately 15 minutes before radiofrequency ablation begins and continue for approximately 30 minutes.
  5% Dextrose Solution: Single 30 minute intravenous infusion
Period: Overall Study
Arm/Group | ThermoDox + RFA | Sham + RFA
Started | 354 | 347
Completed | 244 | 245
Not Completed | 110 | 102

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ThermoDox + RFA | Sham + RFA | Total
Number analyzed (Participants) | 354 | 347 | 701
Age, Customized [Number; unit: participants]
  <40 | 7 | 10 | 17
  40-<45 | 13 | 14 | 27
  45-<50 | 18 | 25 | 43
  50-<55 | 42 | 44 | 86
  55-<60 | 57 | 50 | 107
  60-<65 | 65 | 64 | 129
  65-<70 | 44 | 45 | 89
  70-<75 | 51 | 42 | 93
  75-<80 | 33 | 34 | 67
  80-<85 | 19 | 13 | 32
  85+ | 2 | 4 | 6
  Missing | 3 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 84 | 171
  Male | 267 | 263 | 530
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 42 | 26 | 68
  Japanese | 8 | 11 | 19
  Korean | 83 | 91 | 174
  Taiwanese | 66 | 62 | 128
  Chinese | 115 | 125 | 240
  Other | 40 | 32 | 72
Region of Enrollment [Number; unit: participants]
  United States | 10 | 5 | 15
  Philippines | 18 | 21 | 39
  Taiwan | 68 | 63 | 131
  Hong Kong | 6 | 9 | 15
  Canada | 5 | 10 | 15
  Thailand | 16 | 8 | 24
  Malaysia | 7 | 6 | 13
  Japan | 8 | 10 | 18
  Italy | 32 | 17 | 49
  China | 104 | 104 | 208
  Korea, Republic of | 82 | 92 | 174

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival Will be Measured From the Date of Randomization to the First Date on Which One of the Following Occurs. o Local Recurrence o Any New Distant Intrahepatic HCC Tumor o Any New Extrahepatic HCC Tumor o Death From Any Cause
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: Time to Progression (months)
Arm/Group | ThermoDox + RFA | Sham + RFA
Number analyzed (Participants) | 354 | 347
Time to Progression (months) | 13.97 [11.47 to 19.26] | 13.87 [11.14 to 16.69]

2. Secondary Outcome: Overall Survival as Measured by Time From Randomization to Death or the End of the Study.
Time Frame: 3 years
Measure: Number; unit: Participants (Deaths)
Arm/Group | ThermoDox + RFA | Sham + RFA
Number analyzed (Participants) | 354 | 347
Participants (Deaths) | 189 | 188

3. Secondary Outcome: Number of Participants With Definite Worsening as Per Patient-Reported Outcomes
Description: Number of participants with significant symptom deterioration, defined as greater than or equal to 4-point increase from baseline in the eight-item Functional Assessment of Cancer Therapy-Hepatobiliary Symptom Index.
Time Frame: 3 years
Population: Intent-to-treat (ITT) population
Measure: Number; unit: participants
Arm/Group | ThermoDox + RFA | Sham + RFA
Number analyzed (Participants) | 354 | 347
participants | 53 | 60

4. Secondary Outcome: Number of Participants With Local Recurrence
Description: Number of participants with local progression in the intent-to-treat (ITT) population.
Time Frame: 3 years
Population: Intent-to-treat (ITT) population
Measure: Number; unit: participants
Arm/Group | ThermoDox + RFA | Sham + RFA
Number analyzed (Participants) | 354 | 347
participants | 58 | 55

5. Secondary Outcome: Evaluation of Safety
Time Frame: 3 years
Population: Incidence of treatment-related adverse events (≥ 5% of patients in either group; safety population)
Measure: Number; unit: percentage of overall incidence
Arm/Group | ThermoDox + RFA | Sham + RFA
Number analyzed (Participants) | 343 | 344
percentage of overall incidence | 83 | 35

ADVERSE EVENTS:
Arm/Group | ThermoDox + RFA | Sham + RFA
Serious Adverse Events (participants affected / at risk) | 118/343 | 37/334
Other Adverse Events (participants affected / at risk) | 327/343 | 301/334
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ThermoDox + RFA (N=343) | Sham + RFA (N=334)
Neutropenia (Blood and lymphatic system disorders) | 56 | 0
Leukopenia (Blood and lymphatic system disorders) | 19 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 9 | 0
Pancytopenia (Blood and lymphatic system disorders) | 3 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Bone Marrow Failure (Blood and lymphatic system disorders) | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 2
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 3
Oesophageal Varices Haemorrhage (Gastrointestinal disorders) | 1 | 2
Ascites (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Ileus (Gastrointestinal disorders) | 0 | 2
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Duodenal Ulcer (Gastrointestinal disorders) | 1 | 0
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric Varices Haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0
Large Intestine Perforation (Gastrointestinal disorders) | 1 | 0
Localised Intraabdominal Fluid Collection (Gastrointestinal disorders) | 0 | 1
Mesenteric Vein Thrombosis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Peritoneal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Portal Hypertensive Gastropathy (Gastrointestinal disorders) | 0 | 1
Stress Ulcer (Gastrointestinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 2
Cellulitis (Infections and infestations) | 2 | 0
Liver Abscess (Infections and infestations) | 2 | 0
Neutropenic Sepsis (Infections and infestations) | 2 | 0
Peritonitis Bacterial (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 1 | 1
Septic Shock (Infections and infestations) | 1 | 1
Abdominal Infection (Infections and infestations) | 0 | 1
Anal Abscess (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Furuncle (Infections and infestations) | 1 | 0
Gastritis Viral (Infections and infestations) | 1 | 0
Infected Cyst (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Salmonella Sepsis (Infections and infestations) | 1 | 0
Wound Infection Staphylococcal (Infections and infestations) | 0 | 1
Hepatic Rupture (Injury, poisoning and procedural complications) | 3 | 0
Post Procedural Complication (Injury, poisoning and procedural complications) | 1 | 2
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 2 | 1
Procedural Pain (Injury, poisoning and procedural complications) | 1 | 1
Wound Complication (Injury, poisoning and procedural complications) | 1 | 1
Biloma (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Hepatic Function Abnormal (Injury, poisoning and procedural complications) | 1 | 0
Hypotension (Injury, poisoning and procedural complications) | 0 | 1
Puncture Site Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Wound Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Neutrophil Count Decreased (Investigations) | 9 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 0
Blood Bilirubin Increased (Investigations) | 1 | 0
Haemoglobin Decreased (Investigations) | 1 | 0
Platelet Count Decreased (Investigations) | 1 | 0
White Blood Cell Count Decreased (Investigations) | 1 | 0
Hepatic Function Abnormal (Hepatobiliary disorders) | 2 | 1
Jaundice Cholestatic (Hepatobiliary disorders) | 0 | 2
Bile Duct Stone (Hepatobiliary disorders) | 0 | 1
Hepatic Failure (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Liver Disorder (Hepatobiliary disorders) | 1 | 0
Liver Injury (Hepatobiliary disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 2
Multi-organ Failure (General disorders) | 0 | 2
Asthenia (General disorders) | 0 | 1
Hyperpyrexia (General disorders) | 1 | 0
Oedema Peripheral (General disorders) | 1 | 0
Hepatic encephalopthy (Nervous system disorders) | 1 | 1
Cerebral Ischaemia (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Depressed Level of Consciousness (Nervous system disorders) | 1 | 0
Haemorrhagic Stroke (Nervous system disorders) | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 2 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic Acidosis (Metabolism and nutrition disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 2 | 0
Cardiac Failure (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Myocardial Rupture (Cardiac disorders) | 0 | 1
Pericardial Effusion (Cardiac disorders) | 0 | 1
Acute Prerenal Failure (Renal and urinary disorders) | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 | 0
Urethral Stenosis (Renal and urinary disorders) | 1 | 0
Delirium Tremens (Psychiatric disorders) | 1 | 0
Mood Altered (Psychiatric disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Shock Haemorrhagic (Vascular disorders) | 0 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Tumour Thrombosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Biliary Drainage (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ThermoDox + RFA (N=343) | Sham + RFA (N=334)
Hypertension (Vascular disorders) | 18 | 17
Haematuria (Renal and urinary disorders) | 13 | 23
Decreased Appetite (Metabolism and nutrition disorders) | 32 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 26 | 49
Procedural Pain (Injury, poisoning and procedural complications) | 28 | 39
Wound Complication (Injury, poisoning and procedural complications) | 33 | 33
Alopecia (Skin and subcutaneous tissue disorders) | 173 | 2
Neutropenia (Blood and lymphatic system disorders) | 87 | 6
Leukopenia (Blood and lymphatic system disorders) | 73 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 18 | 2
Pyrexia (General disorders) | 56 | 98
Fatigue (General disorders) | 20 | 14
Aspartate Aminotransferase Increased (Investigations) | 70 | 70
Alanine Aminotransferase Increased (Investigations) | 61 | 62
Blood Bilirubin Increased (Investigations) | 29 | 39
White Blood Cell Count Decreased (Investigations) | 48 | 12
Neutrophil Count Decreased (Investigations) | 38 | 9
Platelet Count Decreased (Investigations) | 20 | 20
Blood Lactate Dehydrogenase Increased (Investigations) | 19 | 17
Neutrophil Count Increased (Investigations) | 24 | 8
White Blood Cell Count Increased (Investigations) | 24 | 5
Abdominal Pain (Gastrointestinal disorders) | 50 | 62
Nausea (Gastrointestinal disorders) | 53 | 43
Abdominal Pain Upper (Gastrointestinal disorders) | 44 | 44
Vomiting (Gastrointestinal disorders) | 35 | 28
Constipation (Gastrointestinal disorders) | 21 | 15
Abdominal Distension (Gastrointestinal disorders) | 15 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less